CLINICAL TRIAL: NCT03847701
Title: Cardio-metabolic and Inflammatory Impact of Starch Digestibility in Type 2 Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other); Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KBE045
Record Dates: First submitted 2019-01-30; First posted 2019-02-20 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Type2 Diabetes
Keywords: Slowly Digestible Starch; SDS; Type 2 diabetes; T2D; Glycemic response; Continuous Glucose Monitoring System; CGMS; Diet; MAGE; Mean Amplitude of Glucose Excursion
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Each participant will be allocated to an intervention arm in a parallel design for 3 months of intervention
Who Masked: Participant, Outcomes Assessor
Masking Description: Each diet will be labelled "Diet A" or "Diet B"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High in SDS (Active Comparator): Balanced diet high in Slowly Digestible Starch
  Interventions: Other: Balanced diet high in Slowly Digestible Starch
- Low in SDS (Placebo Comparator): Balanced diet low in Slowly Digestible Starch
  Interventions: Other: Balanced diet low in Slowly Digestible Starch

INTERVENTIONS:
Other: Balanced diet high in Slowly Digestible Starch — The carbohydrates present in high Slowly Digestible Starch diet were selected according to the general recommendations made for diabetics and according to their SDS content. The diet will be consumed during three months.
  Other Names: Diet A; H-SDS
  Arms: High in SDS
Other: Balanced diet low in Slowly Digestible Starch — The carbohydrates present in low-Slowly Digestible Starch diet were selected according to the general recommendations made for diabetics and according to their SDS content. The diet will be consumed during three months.
  Other Names: Diet B; L-SDS
  Arms: Low in SDS

SUMMARY:
This is a monocentric, randomized, single-blind and controlled study with a parallel design (2 arms). The research hypothesis is that the diet high in Slow Digestible Starch (SDS) content (H-SDS) will lower the daylong glycemic response and improve the glycemic control just as metabolic, inflammatory, cardiovascular and oxidative stress parameters in patients with type 2 diabetes (T2D) compared to the diet low in SDS content (L-SDS). The hypothesis is that these differences in glycemic response and in metabolic, inflammatory, cardiovascular and oxidative stress parameters response can be observed after 3 months of diet.

DETAILED DESCRIPTION:
This is a monocentric, randomized, single-blind and controlled study with a parallel design (2 arms). The research hypothesis is that the diet high in Slow Digestible Starch (SDS) content (H-SDS) will lower the daylong glycemic response and improve the glycemic control just as metabolic, inflammatory, cardiovascular and oxidative stress parameters in patients with type 2 diabetes (T2D) compared to the diet low in SDS content (L-SDS). The hypothesis is that these differences in glycemic response and in metabolic, inflammatory, cardiovascular and oxidative stress parameters response can be observed after 3 months of diet.

80 patients with type 2 diabetes will be recruited.

Subjects will have 11 visits:

V0 = selection visit: check whether the patients fulfill inclusion and exclusion criteria for the study.

Visit V1 = CGMS insertion on usual lifestyle without any changes in his/her diet. This is the Run-in period.

Visit V2 (6 days +/- 1 day) = CGMS removal and randomization according to sex, HbA1c and MAGE.

Visit V3 = first metabolic day: medical check-up, dietary interview, indirect calorimetry, impedancemetry measurements and FlexMeal challenge test with 5h follow up (blood samples). CGMS insertion with detailed dietetic instructions according to their allocated group (adapted food provisions).

Visit V4 (6 days +/- 1 day) = CGMS removal. Arterial Endothelial Function (AEF) measurement. Adapted food provisions.

Visit V5 = Adapted food provisions.

Visit V6 = medical check-up, dietary interview, CGMS insertion and baseline blood measurements. Adapted food provisions.

Visit V7 (6 days +/- 1 day) = CGMS removal. Arterial Endothelial Function (AEF) measurement. Adapted food provisions.

Visit V8 = Adapted food provisions.

Visit V9 = CGMS insertion. Arterial Endothelial Function (AEF) measurement. Adapted food provisions.

Visit V10 (6 days +/- 1 day) = second metabolic day: medical check-up, dietary interview, indirect calorimetry, impedancemetry measurements and FlexMeal challenge test with 5h follow up (blood samples). CGMS removal. Feedback questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patient able to understand the study information and providing written consent for his/her participation to the study
* Male or female
* Patient undergoing medical examination during the selection visit
* Patient aged between 18 and 75 years old (bounds included)
* T2D volunteer with HbA1c between 7% and 8,5% without signs of insulinopenia according to the investigator
* Patient with BMI ranging between 25 and 40 kg/m2 (bounds included)
* Patient with stable body weight over the past three months (+/- 5 % of body weight)
* Patient accepting to change its diet for three months
* Patient not suffering from food intolerance or allergy
* Patient regularly consuming products proposed in the study
* Patient agreeing to consume 3 main meals per day without extra-prandial carbohydrates intakes
* Sedentary behavior or stable predicted physical activity during the study
* Patient not presenting any disease during the medical examination / interview which could interfere with the results of the study according to the investigator
* Patient covered by health insurance
* Patient accepting to have short nails on his/her 2 forefingers

Exclusion Criteria:

* Patient under legal protection measure
* Patient deprived of liberty by a court or an administrative decision
* Patient currently participating in another study or being in the exclusion period of another study
* Volunteer that exceed the financial compensation allowed per year for participating in research programs
* Gamma-GT > 2.5 times above the norm (>160 UI/L)
* ASAT > 2.5 times above the norm (>85 UI/L)
* ALAT > 2.5 times above the norm (>137.5 UI/L)
* Triglycerides > 4 g/L
* LDL-cholesterol > 1.90 g/L
* CRP > 15 mg/L
* Hemoglobin < 120 mg/dL
* eGRF (estimated glomerular filtration rate) < 45 ml/min
* Other biological abnormality with clinical significant relevance according to the investigator
* Patient with type 1 diabetes, post pancreatectomy or post transplant diabetes, MODY diabetes, mitochondrial diabetes, iatrogenic diabetes
* T2D volunteer with any other anti-diabetic treatment other than metformin: insulin therapy, GLP-1 analogues, acarbose, sulphonylureas, repaglinide, SGLT2 agonists,…
* Patient consuming in the two previous months regularly corticoids, beta-blocking drugs or immunosuppressing drugs
* Patient with hemoglobin pathology
* Patient with medical history of hemoglobinopathies (thalassemia, drepanocytosis…)
* Patient with past bariatric surgery
* Patient with medical history of endocrine diseases who may interfere with glucose metabolism according to the investigator (such as hyperthyroidism, acromegaly, hypercorticism…)
* Patient treated with anticoagulants
* Patient with a pace-maker
* Uncontrolled high blood pressure defined by Systolic blood pressure > 150 mmHg or Diastolic blood pressure > 100 mmHg
* Evidence of any other unstable or untreated clinically significant immunological, neoplasic, endocrine, haematological, gastrointestinal, hepatic, neurological or psychiatric abnormalities or medical disease with clinical significant relevance according to the investigator
* Pregnant women or willing to become pregnant or lactating women
* Women of childbearing age without an efficient contraceptive method according to the investigator
* Patient under a restrictive diet or with a planned weight loss program during the study
* Patient with severe eating disorders (e.g. anorexia nervosa, binge eating disorder and bulimia) according to the investigator
* Patient without stable dietary habits or with specific diet (vegetarian, vegan, gluten-free…) according to the investigator
* Patient who smokes more than 5 cigarettes per day
* Patient regularly consuming more than 20 g/day of alcohol. Consumption of more than 3 alcoholic beverages per day is recognized as excessive. An alcoholic beverage is: 30 mL of spirituous, 120 mL of wine or 330 mL of beer
* Patient regularly consuming recreational drugs
* Adhesive plaster skin allergy
* Claustrophobic patient
* Patient willing to take the plane during the CGMS periods

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
MAGE comparison following 3 months of intake of a diet either high or low in SDS | Minimum 3 days to a maximum of 6 days of CGMS record
  Mean Amplitude of Glycemic Excursions (MAGE) from CGMS glycaemia

SECONDARY OUTCOMES:
Glycemia iAUC characterisation of a standard challenge test (FlexMeal) during the first metabolic day | 5 hours post standard challenge test during visit 3
  Glycemia iAUC
Insulin iAUC characterisation of a standard challenge test (FlexMeal) during the first metabolic day | 5 hours post standard challenge test during visit 3
  Insulin iAUC
GLP1 iAUC characterisation of a standard challenge test (FlexMeal) during the first metabolic day | 5 hours post standard challenge test during visit 3
  GLP1 iAUC
Inflammatory status comparison during the first metabolic day : CRPus concentration | At a basal state during visit 3
  CRPus
Inflammatory impacts characterisation of a standard challenge test (FlexMeal) during the first metabolic day : TNFa iAUC | 5 hours post standard challenge test during visit 3
  TNFa iAUC
Inflammatory impacts characterisation of a standard challenge test (FlexMeal) during the first metabolic day : IL6 iAUC | 5 hours post standard challenge test during visit 3
  IL6 iAUC
Inflammatory impacts characterisation of a standard challenge test (FlexMeal) during the first metabolic day : IL1Ra iAUC | 5 hours post standard challenge test during visit 3
  IL1Ra iAUC
Inflammatory impacts characterisation of a standard challenge test (FlexMeal) during the first metabolic day : IL18 iAUC | 5 hours post standard challenge test during visit 3
  IL18 iAUC
Glycemic impacts comparison following the intake of a diet either high or low in SDS during the time course of the study | At a basal state during visit 3, visit 6 and visit 10
  Glycemia concentration
Insulinemic impacts comparison following the intake of a diet either high or low in SDS during the time course of the study | At a basal state during visit 3, visit 6 and visit 10
  Insulin concentration
Inflammatory impacts comparison following the intake of a diet either high or low in SDS during the time course of the study : CRPus concentration | At a basal state during visit 3, visit 6 and visit 10
  CRPus concentration
Inflammatory impacts comparison following the intake of a diet either high or low in SDS during the time course of the study : TNFa concentration | At a basal state during visit 3, visit 6 and visit 10
  TNFa concentration
Inflammatory impacts comparison following the intake of a diet either high or low in SDS during the time course of the study : IL6 concentration | At a basal state during visit 3, visit 6 and visit 10
  IL6 concentration
Inflammatory impacts comparison following the intake of a diet either high or low in SDS during the time course of the study : IL1Ra concentration | At a basal state during visit V3, V6 and V10
  IL1Ra concentration
Inflammatory impacts comparison following the intake of a diet either high or low in SDS during the time course of the study : IL18 concentration | At a basal state during visit 3, visit 6 and visit 10
  IL18 concentration
Oxidative Stress comparison following the intake of a diet either high or low in SDS during the time course of the study : MDA concentration | At a basal state during visit 3, visit 6 and visit 10
  Malonaldehyde : MDA concentration
Oxidative Stress comparison following the intake of a diet either high or low in SDS during the time course of the study : Urinary isoprostanes concentration | At a basal state during visit 3, visit 6 and visit 10
  Urinary isoprostanes concentration
Cardiovascular risk markers comparison following the intake of a diet either high or low in SDS during the time course of the study : MCP1 concentration | At a basal state during visit 3, visit 6 and visit 10
  MCP1 concentration
Cardiovascular risk markers comparison following the intake of a diet either high or low in SDS during the time course of the study : sICAM concentration | At a basal state during visit 3, visit 6 and visit 10
  sICAM concentration
Cardiovascular risk markers comparison following the intake of a diet either high or low in SDS during the time course of the study : sVCAM concentration | At a basal state during visit 3, visit 6 and visit 10
  sVCAM concentration
Glycemic impacts characterisation of a standard challenge test (FlexMeal) during the second metabolic day | 5 hours post standard challenge test during visit 10
  Glycemia iAUC
Insulinemic impacts characterisation of a standard challenge test (FlexMeal) during the second metabolic day | 5 hours post standard challenge test during visit 10
  Insulin iAUC
GLP1 iAUC characterisation of a standard challenge test (FlexMeal) during the second metabolic day | 5 hours post standard challenge test during visit 10
  GLP1 iAUC
Inflammatory impacts comparison following 3 months of intake of a diet either high or low in SDS : CRPus concentration | At a basal state during visit 10
  CRPus concentration
Inflammatory impacts characterisation of a standard challenge test (FlexMeal) during the second metabolic day : TNFa iAUC | 5 hours post standard challenge test during visit 10
  TNFa iAUC
Inflammatory impacts characterisation of a standard challenge test (FlexMeal) during the second metabolic day : IL6 iAUC | 5 hours post standard challenge test during visit 10
  IL6 iAUC
Inflammatory impacts characterisation of a standard challenge test (FlexMeal) during the second metabolic day : IL1Ra iAUC | 5 hours post standard challenge test during visit 10
  IL1Ra iAUC
Inflammatory impacts characterisation of a standard challenge test (FlexMeal) during the second metabolic day : IL18 iAUC | 5 hours post standard challenge test during visit 10
  IL18 iAUC
Cardiovascular risk markers characterisation following the intake of a diet either high or low in SDS : MCP1 concentration | After 3 months consumption of the diet
  MCP1 concentration
Cardiovascular risk markers characterisation following the intake of a diet either high or low in SDS : sICAM concentration | After 3 months consumption of the diet
  sICAM concentration
Cardiovascular risk markers characterisation following the intake of a diet either high or low in SDS : sVCAM concentration | After 3 months consumption of the diet
  sVCAM concentration
Oxydative stress characterisation following the intake of a diet either high or low in SDS : MDA concentration | After 3 months consumption of the diet
  Malonaldehyde : MDA concentration
Oxydative stress characterisation following the intake of a diet either high or low in SDS : Urinary isoprostanes concentration | After 3 months consumption of the diet
  Urinary isoprostanes concentration
Glycemic profile parameters following the intake of a diet either high or low in SDS during the time course of the study : MAGE | minimum 3 days to a maximum of 6 days of CGMS record
  Mean Amplitude of Glycemic Excursions (MAGE) from CGMS glycaemia
Glycemic profile parameters following the 3 months consumption of a diet either high or low in SDS : MAGE | after 3 months consumption of the diet, CGMS record for a minimum of 3 days to a maximum of 6 days
  Mean Amplitude of Glycemic Excursions (MAGE) from CGMS glycaemia
Glycemic profile parameters following the intake of a diet either high or low in SDS during the time course of the study : TIR | minimum 3 days to a maximum of 6 days of CGMS record
  Time In Range (TIR) from CGMS glycaemia
Glycemic profile parameters following the 3 months consumption of a diet either high or low in SDS : TIR | after 3 months consumption of the diet, CGMS record for a minimum of 3 days to a maximum of 6 days
  Time In Range (TIR) from CGMS glycaemia
Glycemic profile parameters following the intake of a diet either high or low in SDS during the time course of the study : CV | minimum 3 days to a maximum of 6 days of CGMS record
  Coefficient of Variation (CV) from CGMS glycaemia
Glycemic profile parameters following the 3 months consumption of a diet either high or low in SDS : CV | after 3 months consumption of the diet, CGMS record for a minimum of 3 days to a maximum of 6 days
  Coefficient of Variation (CV) from CGMS glycaemia
Glycemic profile parameters following the intake of a diet either high or low in SDS during the time course of the study : SD | minimum 3 days to a maximum of 6 days of CGMS record
  Standard Deviation (SD) from CGMS glycaemia
Glycemic profile parameters following the 3 months consumption of a diet either high or low in SDS : SD | after 3 months consumption of the diet, CGMS record for a minimum of 3 days to a maximum of 6 days
  Standard Deviation (SD) from CGMS glycaemia
Glycemic profile parameters following the intake of a diet either high or low in SDS during the time course of the study : MIME | minimum 3 days to a maximum of 6 days of CGMS record
  Mean Indices of Meal Excursions (MIME) from CGMS glycaemia
Glycemic profile parameters following the 3 months consumption of a diet either high or low in SDS : MIME | after 3 months consumption of the diet, CGMS record for a minimum of 3 days to a maximum of 6 days
  Mean Indices of Meal Excursions (MIME) from CGMS glycaemia
Glycemic profile parameters following the intake of a diet either high or low in SDS during the time course of the study : MODD | minimum 3 days to a maximum of 6 days of CGMS record
  Mean Of Daily Differences (MODD) from CGMS glycaemia
Glycemic profile parameters following the 3 months consumption of a diet either high or low in SDS : MODD | after 3 months consumption of the diet, CGMS record for a minimum of 3 days to a maximum of 6 days
  Mean Of Daily Differences (MODD) from CGMS glycaemia
Glycemic profile parameters following the intake of a diet either high or low in SDS during the time course of the study : CONGA | minimum 3 days to a maximum of 6 days of CGMS record
  Continuous Overall Net Glycemic Action (CONGA) from CGMS glycaemia
Glycemic profile parameters following the 3 months consumption of a diet either high or low in SDS : CONGA | after 3 months consumption of the diet, CGMS record for a minimum of 3 days to a maximum of 6 days
  Continuous Overall Net Glycemic Action (CONGA) from CGMS glycaemia
Glycemic profile parameters following the intake of a diet either high or low in SDS during the time course of the study : ADRR | minimum 3 days to a maximum of 6 days of CGMS record
  Average Daily Risk Range (ADRR) from CGMS glycaemia
Glycemic profile parameters following the 3 months consumption of a diet either high or low in SDS : ADRR | after 3 months consumption of the diet, CGMS record for a minimum of 3 days to a maximum of 6 days
  Average Daily Risk Range (ADRR) from CGMS glycaemia
Glycemic profile parameters following the intake of a diet either high or low in SDS during the time course of the study : LGBI | minimum 3 days to a maximum of 6 days of CGMS record
  Low Blood Glucose Index (LGBI) from CGMS glycaemia
Glycemic profile parameters following the 3 months consumption of a diet either high or low in SDS : LGBI | after 3 months consumption of the diet, CGMS record for a minimum of 3 days to a maximum of 6 days
  Low Blood Glucose Index (LGBI) from CGMS glycaemia
Glycemic profile parameters following the intake of a diet either high or low in SDS during the time course of the study : HGBI | minimum 3 days to a maximum of 6 days of CGMS record
  High Blood Glucose Index (HGBI) from CGMS glycaemia
Glycemic profile parameters following the 3 months consumption of a diet either high or low in SDS : HGBI | after 3 months consumption of the diet, CGMS record for a minimum of 3 days to a maximum of 6 days
  High Blood Glucose Index (HGBI) from CGMS glycaemia
Mean daylong incremental Area Under the Curve (iAUC), measured by CGMS, following the intake of a diet either high or low in SDS during the time course of the study | from 0 min to 360 min postprandial during the CGMS record periods (from visit 3 to visit 4, from visit 6 to visit 7 and from visit 9 to visit 10)
  The iAUC will be calculated using the trapezoid rule. The iAUC includes all area below the curve and above the fasting concentration, with any area beneath fasting being ignored.
Mean daylong total Area Under the Curve (tAUC), measured by CGMS, following the intake of a diet either high or low in SDS during the time course of the study | from 0 min to 360 min postprandial during the CGMS record periods (from visit 3 to visit 4, from visit 6 to visit 7 and from visit 9 to visit 10)
  The tAUC will be calculated using the trapezoid rule.
Compare diabetes follow-up markers during the first metabolic day : HbA1c | At the basal state during visit 3
  Hba1c concentration
Compare diabetes follow-up markers following the intake of a diet either high or low in SDS during the time course of the study : HbA1c concentration | At a basal state, during visit 3, visit 6 and visit 10
  Hba1c
Compare diabetes follow-up markers following the 3 months consumption of a diet either high or low in SDS : HbA1c concentration | After 3 months consumption of the diet, at the basal state
  Hba1c
Compare Diabetes follow-up markers during the first metabolic day : Fructosamine concentration | At the basal state during visit 3
  Fructosamine
Compare Diabetes follow-up markers following the intake of a diet either high or low in SDS during the time course of the study : fructosamine concentration | At a basal state, during visit 3, visit 6 and visit 10
  Fructosamine
Compare Diabetes follow-up markers following the 3 months consumption of a diet either high or low in SDS : Fructosamine concentration | After 3 months consumption of the diet, at the basal state
  Fructosamine
Compare Diabetes follow-up markers during the first metabolic day : Glycated Albumin concentration | At the basal state during visit 3
  Glycated albumin
Compare Diabetes follow-up markers following the intake of a diet either high or low in SDS during the time course of the study : glycated albumin concentration | At a basal state, during visit 3, visit 6 and visit 10
  Glycated albumin
Compare Diabetes follow-up markers following the 3 months consumption of a diet either high or low in SDS : Glycated Albumin concentration | After 3 months consumption of the diet, at the basal state
  Glycated albumin
Arterial Endothelial Function characterisation following the intake of a diet either high or low in SDS during the time course of the study : RHI | At a basal state during visit 4, visit 7 and visit 9
  Reactive Hyperemia (RHI)
Arterial Endothelial Function characterisation following the intake of a diet either high or low in SDS during the time course of the study : AI | At a basal state during visit 4, visit 7 and visit 9
  Augmentation Index (AI)
Arterial Endothelial Function characterisation following the intake of a diet either high or low in SDS during the time course of the study : HRV | At a basal state during visit 4, visit 7 and visit 9
  Heart Rate Variability (HRV)
Anthropometry parameters characterisation during the first metabolic day : height | At baseline during visit 3
  Height
Anthropometry parameters characterisation during the first metabolic day : body weight | At baseline during visit 3
  body weight
Anthropometry parameters characterisation during the first metabolic day : waist circumference | At baseline during visit 3
  waist circumference
Anthropometry parameters characterisation during the first metabolic day : hip circumference | At baseline during visit 3
  hip circumference
Anthropometry parameters characterisation following the intake of a diet either high or low in SDS during the time course of the study : height | At baseline during visit 3, visit 6 and visit 10
  Height
Anthropometry parameters characterisation following the intake of a diet either high or low in SDS during the time course of the study : body weight | At baseline during visit 3, visit 6 and visit 10
  body weight
Anthropometry parameters characterisation following the intake of a diet either high or low in SDS during the time course of the study : waist circumference | At baseline during visit 3, visit 6 and visit 10
  waist circumference
Anthropometry parameters characterisation following the intake of a diet either high or low in SDS during the time course of the study : hip circumference | At baseline during visit 3, visit 6 and visit 10
  hip circumference
Anthropometry parameters characterisation following the 3 months consumption of a diet either high or low in SDS : height | At baseline during visit 10
  Height
Anthropometry parameters characterisation following the 3 months consumption of a diet either high or low in SDS : body weight | At baseline during visit 10
  body weight
Anthropometry parameters characterisation following the 3 months consumption of a diet either high or low in SDS : waist circumference | At baseline during visit 10
  waist circumference
Anthropometry parameters characterisation following the 3 months consumption of a diet either high or low in SDS : hip circumference | At baseline during visit 10
  hip circumference
Body composition parameters characterisation during the first metabolic day: total body water | At baseline during visit 3
  Total body water measured by bioimpedancemetry
Body composition parameters characterisation during the first metabolic day: body fat | At baseline during visit 3
  Body fat measured by bioimpedancemetry
Body composition parameters characterisation during the first metabolic day: lean mass. | At baseline during visit 3
  Lean mass measured by bioimpedancemetry
Body composition parameters characterisation following the 3 months consumption of a diet either high or low in SDS : total body water | At baseline during visit 10
  Total body water measured by bioimpedancemetry
Body composition parameters characterisation following the 3 months consumption of a diet either high or low in SDS : body fat | At baseline during visit 10
  Body fat measured by bioimpedancemetry
Body composition parameters characterisation following the 3 months consumption of a diet either high or low in SDS : lean mass | At baseline during visit 10
  Lean mass measured by bioimpedancemetry
Resting energy metabolism profile during the first metabolic day: Resting Metabolism Rate | At baseline during visit 3
  Resting Metabolism Rate (RMR)
Resting energy metabolism profile following the 3 months consumption of a diet either high or low in SDS : Resting Metabolism Rate | At baseline during visit 10
  Resting Metabolism Rate (RMR)
Diabetic glycemic variability characterisation following the 3 months consumption of a diet either high or low in SDS | after 3 months consumption of the diet, CGMS record for a minimum of 3 days to a maximum of 6 days
  Percent of subjects reaching the target for HbA1C, TIR and CV
Level of physical activity characterisation following the intake of a diet either high or low in SDS during the time course of the study : IPAQ | After each CGMS record periods, ie : at visit 4, visit 7 and visit 10
  International Physical Activity Questionnaire (IPAQ)
Characterisation of acceptability to H-SDS diet in free living conditions | After 3 months consumption of the diet, at visit 10
  Feedback questionnaire
Characterisation of the percent of compliance to H-SDS diet in free living conditions | After 3 months consumption of the diet
  Table of compliance in the volunteer's notebook. Subjects will have to fulfill it after each meal during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel DISSE, MD, PhD, Principal Investigator — Centre de Recherche en Nutrition Humaine Rhône-Alpes; Martine LAVILLE, MD, PhD, Study Chair — Centre de Recherche en Nutrition Humaine Rhône-Alpes
Locations (1):
- Centre de Recherche en Nutrition Humaine Rhone-Alpes, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chisbert M, Castell AL, Van Den Berghe L, Breyton AE, Feugier N, Cuerq C, Chikh K, Brack O, Laville M, Goux A, Meynier A, Vinoy S, Nazare JA. Optimizing glycemic variability in type 2 diabetes using simple dietary and culinary recommendations to modulate starch digestibility: a randomized controlled trial. Am J Clin Nutr. 2025 Dec;122(6):1591-1601. doi: 10.1016/j.ajcnut.2025.10.007. Epub 2025 Oct 13. PMID 41092985